CLINICAL TRIAL: NCT07130292
Title: Effects of Abdominal Muscle Strengthening Using Stabilizer Pressure Biofeedback on Menstrual Symptoms and Abdominal Muscle Strength in Young Women With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Abdominal Muscle Strengthening for Menstrual Symptoms in Primary Dysmenorrhea
Acronym: STAMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sanem ŞENER, Assistant Professor, PhD, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZBEU-SPB-PD-2025-01
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Menstrual Pain; Menstrual Disorders; Muscle Strength
Keywords: Primary Dysmenorrhea; Abdominal Muscle Strengthening; Stabilizer Pressure Biofeedback
MeSH Terms: conditions — Dysmenorrhea; Menstruation Disturbances

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups: an intervention group receiving abdominal muscle strengthening and stretching exercises guided by a stabilizer pressure biofeedback device, and a control group receiving no such intervention during the study period. Both groups will be evaluated at baseline, mid-intervention, and post-intervention over an 8-week period.
Who Masked: Outcomes Assessor
Masking Description: This study uses a single-blind design in which the outcomes assessor is unaware of participants' group allocation. Participants and care providers are aware of the assigned interventions, but the assessor responsible for data collection and outcome evaluation remains blinded throughout the trial to reduce measurement bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Abdominal Muscle Strengthening with Stabilizer Pressure Biofeedback (Experimental): Participants perform a structured exercise program targeting lumbar and abdominal muscles, guided by a stabilizer pressure biofeedback device. Sessions are supervised three times per week for 6 weeks (excluding menstruation weeks) and include mobility, stretching, and strengthening exercises to improve abdominal muscle activation and core stability.
  Interventions: Behavioral: Abdominal Muscle Strengthening Exercises with Stabilizer Pressure Biofeedback
- Control - No Abdominal Muscle Strengthening Intervention (No Intervention): Participants receive no abdominal muscle strengthening program during the study period. They continue their usual daily activities without any supervised exercise intervention.

INTERVENTIONS:
Behavioral: Abdominal Muscle Strengthening Exercises with Stabilizer Pressure Biofeedback — A supervised exercise program designed to strengthen abdominal and lumbar muscles, incorporating the use of a stabilizer pressure biofeedback device to enhance activation of deep stabilizing muscles such as the transversus abdominis. The program is delivered three times per week for 6 weeks (excluding menstruation weeks) and includes mobility, stretching, and strengthening exercises.
  Arms: Intervention - Abdominal Muscle Strengthening with Stabilizer Pressure Biofeedback

SUMMARY:
This randomized controlled trial aims to investigate the effects of abdominal muscle strengthening exercises using a stabilizer pressure biofeedback device on menstrual symptoms and abdominal muscle strength in young women with primary dysmenorrhea. Primary dysmenorrhea, characterized by painful menstrual cramps without underlying pelvic pathology, is common among women of reproductive age and can negatively affect quality of life.

In this study, 58 female participants aged 18-25 with regular menstrual cycles and a Visual Analog Scale (VAS) pain score of ≥4 will be randomly assigned to either an intervention group or a control group. The intervention group will perform abdominal strengthening and stretching exercises guided by a stabilizer pressure biofeedback device, three times per week for 6 weeks (excluding menstruation weeks).

The main outcomes include menstrual symptom severity (assessed by the Menstrual Symptom Scale), pain intensity (VAS), and abdominal muscle strength (measured using the stabilizer pressure biofeedback device). The results will help determine whether targeted abdominal muscle training can reduce menstrual symptoms and improve muscle strength in women with primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is one of the most common gynecological problems in women of reproductive age, characterized by spasmodic cramps in the lower abdomen before or during menstruation, without pelvic pathology. The underlying pathophysiology involves increased release of prostaglandin F2α during menstruation, leading to stronger uterine contractions, reduced blood flow, hypoxia, and pain. PD often begins soon after menarche and may be accompanied by nausea, vomiting, diarrhea, fatigue, and sleep disturbances.

Conventional treatment approaches include pharmacological methods such as nonsteroidal anti-inflammatory drugs (NSAIDs) and hormonal contraceptives. However, these treatments may have side effects and limited patient compliance. Non-pharmacological interventions, especially exercise programs, have shown potential in reducing menstrual pain by increasing endorphin release, relaxing uterine muscles, and improving regional blood flow. Strengthening abdominal and core muscles can improve pelvic stability and potentially reduce dysmenorrhea symptoms.

The stabilizer pressure biofeedback unit is a simple, non-invasive device that provides visual feedback during muscle activation, helping to target deep stabilizing muscles such as the transversus abdominis. By enhancing activation capacity, it may improve abdominal muscle strength and reduce menstrual symptoms.

Study Design:

This is a randomized, controlled, single-blind trial. Fifty-eight eligible women aged 18-25 with regular menstrual cycles, a VAS score ≥4, and no diagnosis of secondary dysmenorrhea or other gynecological disorders will be enrolled. Participants will be allocated to the intervention or control group using permuted block randomization. Assessments will be conducted three times: at baseline (first day of the menstrual cycle), mid-intervention (week 3-4), and post-intervention (week 8).

Intervention:

The intervention group will perform a structured exercise program targeting the lumbar and abdominal muscles, supervised three times per week for 6 weeks (excluding menstruation weeks). Exercises will include stretching, mobility, and strengthening activities, with abdominal muscle training guided by a stabilizer pressure biofeedback device. The control group will not receive this intervention during the study period.

Outcome Measures:

Primary outcomes: Menstrual symptom severity (Menstrual Symptom Scale), pain intensity (VAS).

Secondary outcome: Abdominal muscle strength (stabilizer pressure biofeedback).

Significance:

This study will provide evidence on whether non-pharmacological abdominal muscle strengthening using stabilizer pressure biofeedback can reduce menstrual symptoms and improve muscle strength in young women with primary dysmenorrhea. The findings may guide future exercise-based interventions for menstrual pain management.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-25 years
* Regular menstrual cycles
* Diagnosed with primary dysmenorrhea (no secondary dysmenorrhea or other gynecological disorders)
* Menstrual pain intensity ≥ 4 on the Visual Analog Scale (VAS) during the menstrual cycle
* Willingness to participate and ability to provide informed consent

Exclusion Criteria:

* Diagnosis of secondary dysmenorrhea or other gynecological disorders (e.g., endometriosis, adenomyosis, uterine fibroids)
* Current pregnancy or breastfeeding
* History of abdominal or pelvic surgery in the past 6 months
* Current use of hormonal therapy or analgesic medication that could affect menstrual pain assessment
* Participation in regular abdominal or core strengthening exercise programs within the last 3 months
* Any musculoskeletal, neurological, or systemic condition that could interfere with exercise performance or study participation

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-08-13 (Estimated); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Menstrual Symptom Severity | Change from Baseline (Week 0) to Post-intervention (Week 8)
  Change in menstrual symptom severity as assessed by the Menstrual Symptom Scale (MSS). The MSS consists of 22 items scored on a 5-point Likert scale, with higher scores indicating more severe symptoms.
Pain Intensity | Change from Baseline (Week 0) to Post-intervention (Week 8)
  Visual Analog Scale 0-10 cm (0 = no pain, 10 = worst pain). Outcome is mean change from baseline to Week 8.
Abdominal Muscle Activation/Strength (Pressure Biofeedback) | Change from Baseline (Week 0) to Post-intervention (Week 8)
  Abdominal muscle activation measured with a Stabilizer Pressure Biofeedback Unit (mmHg). Lower pressure during correct drawing-in reflects better transversus abdominis activation. Outcome is change from baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Assistant Professor of Physiotherapy, Principal Investigator — Zonguldak Bulent Ecevit University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study protocol and informed consent do not include provisions for public data sharing, and data protection regulations restrict the release of personally identifiable health information.